CLINICAL TRIAL: NCT05340179
Title: Comparison of the Efficacy of Cervical Epidural Steroid Injection and Selective Nerve Root Block in Patients With Cervical Radicular Pain
Brief Title: Efficacy of Cervical Epidural Injection and Selective Nerve Root Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Diskapi Teaching and Research Hospital (Other)
Responsible Party: Principal Investigator, Selin Guven Kose, principal Investigator, Diskapi Teaching and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 131/10
Record Dates: First submitted 2022-04-14; First posted 2022-04-22 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-05

CONDITIONS: Cervical Radiculopathy
MeSH Terms: conditions — Radiculopathy

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interlaminar cervical epidural steroid injection (Active Comparator)
  Interventions: Procedure: Interlaminar cervical epidural injection
- Cervical selective nerve root block (Experimental)
  Interventions: Procedure: Cervical selective nerve root block

INTERVENTIONS:
Procedure: Interlaminar cervical epidural injection — Fluoroscopy-guided interlaminar cervical epidural injection
  Arms: Interlaminar cervical epidural steroid injection
Procedure: Cervical selective nerve root block — Ultrasound-guided cervical selective nerve root block
  Arms: Cervical selective nerve root block

SUMMARY:
Cervical epidural steroid injections are an accepted treatment modality for radicular pain secondary to disc pathology. With the developing ultrasound technology, ultrasound guided cervical selective nerve root block has been successfully used in the treatment of cervical radiculopathy. We aimed to compare the efficacy of cervical interlaminar epidural injections and cervical selective nerve root block.

ELIGIBILITY:
Inclusion Criteria:

* Cervical radicular pain based on history and physical exam
* NRS pain score > 3

Exclusion Criteria:

* Previous spine surgery
* Allergic reactions to drugs used in procedure
* Epidural steroid injection within past 2 years
* Radiculopathy not resulting from disc pathology (e.g. foraminal stenosis or tumor)
* Untreated coagulopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-04-25 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Reduction in pain | Change from baseline pain score to 6months
  Pain assessment will be performed using the Numerical Rating Scale (NRS) score (0 = no pain, 10 = the most severe pain felt).

SECONDARY OUTCOMES:
Neck Disability Index | baseline to 6 months post-procedure

CONTACTS AND LOCATIONS:
Overall Officials: selin guven kose, Principal Investigator — Diskapi Yildirim Beyazit Education and Research Hospital
Locations (1):
- Diskapi Yildirim Beyazit Training and Research Hospital, Ankara, Turkey (Türkiye)